CLINICAL TRIAL: NCT00713830
Title: A Randomized, Double-blind, Placebo-controlled, 2-arm Parallel-group, Multicenter 24-week Study Followed by an Extension Assessing the Efficacy and Safety of AVE0010 on Top of a Sulfonylurea in Patients With Type 2 Diabetes Not Adequately Controlled With Sulfonylurea
Brief Title: GLP-1 Receptor Agonist Lixisenatide in Patients With Type 2 Diabetes for Glycemic Control and Safety Evaluation, on Top of Sulfonylurea
Acronym: GETGOAL-S
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC6015; EudraCT 2007-005881-11
Record Dates: First submitted 2008-07-10; First posted 2008-07-14 (Estimated); Results first posted 2016-12-14 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: hyperglycemia, GLP-1
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia | interventions — lixisenatide; Sulfonylurea Compounds; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lixisenatide (Experimental): 2-step initiation regimen of lixisenatide: 10 microgram (mcg) once daily (QD) for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to the end of treatment.
  Interventions: Drug: Lixisenatide (AVE0010); Device: Pen auto-injector; Drug: Sulfonylurea; Drug: Metformin
- Placebo (Placebo Comparator): 2-step initiation regimen of volume matching placebo: 10 mcg QD for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to the end of treatment.
  Interventions: Drug: Placebo; Device: Pen auto-injector; Drug: Sulfonylurea; Drug: Metformin

INTERVENTIONS:
Drug: Lixisenatide (AVE0010) — Self administered by subcutaneous injections once daily within the hour preceding breakfast.
  Arms: Lixisenatide
Drug: Placebo — Self administered by subcutaneous injections once daily within the hour preceding breakfast.
  Arms: Placebo
Device: Pen auto-injector
  Other Names: OptiClik®
Drug: Sulfonylurea — Sulfonylurea to be continued at maximum effective dose according to local labeling up to end of treatment.
Drug: Metformin — Metformin if given to be continued at stable dose (at least 1.5 gram per day [except at least 0.75 gram per day in Japan and 1.0 gram per day in South Korea]) up to the end of treatment.

SUMMARY:
The purpose of this study is to evaluate the benefits and risks of lixisenatide (AVE0010), in comparison to placebo, as an add-on treatment to sulfonylurea without or with metformin, over a period of 24 weeks of treatment, followed by an extension.

The primary objective is to assess the effects of lixisenatide when added to sulfonylurea with or without metformin on glycemic control in terms of glycosylated hemoglobin (HbA1c) reduction (absolute change) at Week 24.

The secondary objectives are to assess the effects of lixisenatide on percentage of patients reaching HbA1c less than (<) 7 percent (%); percentage of patients reaching HbA1c less than or equal to (<=) 6.5%; body weight; fasting plasma glucose (FPG); beta-cell function assessed by homeostasis model assessment (HOMA) beta; 2-hour postprandial plasma glucose (PPG), glucagon, insulin, proinsulin, and C-peptide after a standardized meal challenge test in a sub-study in all patients in selected centers; to evaluate safety, tolerability, pharmacokinetics (PK) and anti-lixisenatide antibody development.

DETAILED DESCRIPTION:
Patients who complete the 24-week main double-blind treatment would undergo a variable double-blind extension treatment, which ends for all patients at approximately the scheduled date of Week 76 visit (Visit 25) for the last randomized patient.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus, diagnosed for at least 1 year before screening visit, insufficiently controlled with a sulfonylurea alone or a sulfonylurea in association with metformin

Exclusion Criteria:

* HbA1c less than (<) 7% or greater than (>) 10% at screening
* At the time of screening age less than legal age of majority
* Pregnant or breastfeeding women or women of childbearing potential with no effective contraceptive method
* Type 1 diabetes mellitus
* Sulfonylurea less than the maximum effective dose according to local labeling
* Sulfonylurea not at a stable (unchanged) dose for at least 3 months prior to screening
* In case of treatment with metformin in association with sulfonylurea, no stable (unchanged) treatment with metformin of at least 1.5 gram per day (except at least 0.75 gram per day in Japan and at least 1.0 gram per day in South Korea), for at least 3 months prior to screening visit
* FPG at screening >250 milligram per deciliter (mg/dL) (>13.9 millimole per liter [mmol/L])
* History of hypoglycemia unawareness
* Body mass index less than or equal to (<=) 20 kilogram per square meter (kg/m^2)
* Weight change of >5 kg during the 3 months preceding the screening visit
* History of unexplained pancreatitis, chronic pancreatitis, pancreatectomy, stomach/gastric surgery, inflammatory bowel disease
* History of metabolic acidosis, including diabetic ketoacidosis within 1 year prior to screening
* Hemoglobinopathy or hemolytic anemia, receipt of blood or plasma products within 3 months prior to the time of screening
* Within the last 6 months prior to screening, history of myocardial infarction, stroke, or heart failure requiring hospitalization
* Known history of drug or alcohol abuse within 6 months prior to the time of screening
* Cardiovascular, hepatic, neurological, endocrine disease, active malignant tumor or other major systemic disease or patients with short life expectancy making implementation of the protocol or interpretation of the study results difficult, history or presence of clinically significant diabetic retinopathy, history or presence of macular edema likely to require laser treatment within the study period
* Uncontrolled or inadequately controlled hypertension at the time of screening with a resting systolic blood pressure (SBP) or diastolic blood pressure (DBP) >180 millimeter of mercury (mmHg) or >95 mmHg, respectively
* Laboratory findings at the time of screening: aspartate aminotransferase, alanine aminotransferase, or alkaline phosphatase: >2 times upper limit of the normal (ULN) laboratory range; amylase and/or lipase: >3 times ULN; total bilirubin: >1.5 times ULN (except in case of Gilbert's syndrome); hemoglobin <11 gram/deciliter and/or neutrophils <1500 per cubic millimeter (mm^3) and/or platelets <100 000/mm^3; positive test for Hepatitis B surface antigen and/or Hepatitis C antibody
* Any clinically significant abnormality identified on physical examination, laboratory tests or vital signs at the time of screening that in the judgment of the Investigator or any sub investigator precludes safe completion of the study or constrains efficacy assessment
* Patients who are considered by the Investigator or any sub investigator as inappropriate for this study for any reason (for example, impossibility to meet specific protocol requirements, such as scheduled visits, being able to do self-injections, likelihood of requiring treatment during the screening phase and treatment phase with drugs not permitted by the clinical study protocol, Investigator or any sub investigator, pharmacist, study coordinator, other study staff or relative thereof directly involved in the conduct of the protocol)
* Patients with condition/concomitant diseases making them non-evaluable for the efficacy assessment
* Use of oral or injectable antidiabetic or hypoglycemic agents other than sulfonylurea and metformin (for example, alpha glucosidase inhibitor, thiazolidinedione, rimonabant, exenatide, dipeptidyl-peptidase 4 (DPP-4) inhibitors, insulin) within 3 months prior to the time of screening
* Use of systemic glucocorticoids (excluding topical application or inhaled forms) for 1 week or more within 3 months prior to the time of screening
* Use of any investigational drug within 3 months prior to study
* Any previous treatment with lixisenatide (for example, participation in a previous study with lixisenatide)
* Renal impairment defined with serum creatinine >1.4 mg/dL in women and serum creatinine >1.5 mg/dL in men (applicable only for patients with metformin treatment)
* End-stage renal disease as defined by a serum creatinine clearance of <15 milliliter/minute (calculated by the Cockcroft and Gault formula) and/or patients on dialysis (if no treatment with metformin)
* Clinically relevant history of gastrointestinal disease associated with prolonged nausea and vomiting, including, but not limited to gastroparesis and gastroesophageal reflux disease requiring medical treatment, within 6 months prior to the time of screening
* Allergic reaction to any glucagon like peptide-1 (GLP-1) agonist in the past (for example, exenatide, liraglutide) or to metacresol
* Additional exclusion criteria at the end of the run-in phase: informed consent withdrawal; lack of compliance during the single-blind placebo run-in phase (>2 injections missed); and patient with any adverse event which precludes the inclusion in the study, as assessed by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 859 (Actual)
Dates: Start 2008-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (16):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Sofia, Bulgaria
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Cairo, Egypt
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Mumbai, India
- Sanofi-Aventis Administrative Office, Netanya, Israel
- Sanofi-Aventis Administrative Office, Tokyo, Japan
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Seoul, South Korea
- Sanofi-Aventis Administrative Office, Taipei, Taiwan
- Sanofi-Aventis Administrative Office, Bangkok, Thailand
- Sanofi-Aventis Administrative Office, Mégrine, Tunisia
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Rosenstock J, Hanefeld M, Shamanna P, Min KW, Boka G, Miossec P, Zhou T, Muehlen-Bartmer I, Ratner RE. Beneficial effects of once-daily lixisenatide on overall and postprandial glycemic levels without significant excess of hypoglycemia in type 2 diabetes inadequately controlled on a sulfonylurea with or without metformin (GetGoal-S). J Diabetes Complications. 2014 May-Jun;28(3):386-92. doi: 10.1016/j.jdiacomp.2014.01.012. Epub 2014 Jan 28. PMID 24650952
- [Derived] Ahren B, Galstyan G, Gautier JF, Giorgino F, Gomez-Peralta F, Krebs M, Nikonova E, Stager W, Vargas-Uricoechea H. Postprandial Glucagon Reductions Correlate to Reductions in Postprandial Glucose and Glycated Hemoglobin with Lixisenatide Treatment in Type 2 Diabetes Mellitus: A Post Hoc Analysis. Diabetes Ther. 2016 Sep;7(3):583-90. doi: 10.1007/s13300-016-0179-6. Epub 2016 Jun 18. PMID 27319011
- [Derived] Yabe D, Ambos A, Cariou B, Duvnjak L, Evans M, Gonzalez-Galvez G, Lin J, Nikonova EV, de Pablos-Velasco P, Yale JF, Ahren B. Efficacy of lixisenatide in patients with type 2 diabetes: A post hoc analysis of patients with diverse beta-cell function in the GetGoal-M and GetGoal-S trials. J Diabetes Complications. 2016 Sep-Oct;30(7):1385-92. doi: 10.1016/j.jdiacomp.2016.05.018. Epub 2016 May 24. PMID 27267268
- [Derived] Seino H, Onishi Y, Naito Y, Komatsu M. Lixisenatide improves glycemic outcomes of Japanese patients with type 2 diabetes: a meta-analysis. Diabetol Metab Syndr. 2016 Jun 1;8:36. doi: 10.1186/s13098-016-0151-7. eCollection 2016. PMID 27252787

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 136 centers in 16 countries between July 08, 2008 and January 14, 2011. The overall duration of treatment was at least 76 weeks (24 weeks main double-blind treatment; variable double-blind extension treatment).
Pre-assignment Details: A total of 1438 participants were screened of which 579 (40.3%) were screen failures; main reason for screen failure was glycosylated hemoglobin (HbA1c) values being out of the defined protocol range (greater than or equal to 7% and less than or equal to 10%). A total of 859 participants were randomized.
Groups:
- Placebo: 2-step initiation regimen of volume matching placebo: 10 microgram (mcg) once daily (QD) subcutaneously for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to the end of treatment.
- Lixisenatide: 2-step initiation regimen of lixisenatide: 10 mcg QD subcutaneously for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to the end of treatment.
Period: Overall Study
Arm/Group | Placebo | Lixisenatide
Started | 286 (Randomized.) | 573
Modified Intent-to-Treat(mITT)Population | 286 (All patients who received at least 1 dose;had baseline,at least 1 post-baseline efficacy assessment.) | 570
Safety Population | 285 (All patients who were exposed to at least 1 dose, regardless of amount of treatment administered.) | 574 (1 patient randomized to placebo received Lixisenatide (at least one dose))
Subgroup for Standardized Meal Test | 155 (Patients at selected sites where standardized meal challenge test was performed.) | 313
Completed | 204 | 396
Not Completed | 82 | 177
Not completed — Adverse Event | 23 | 71
Not completed — Lack of Efficacy | 24 | 16
Not completed — Lost to Follow-up | 2 | 9
Not completed — Withdrawal by Subject | 13 | 23
Not completed — Poor Compliance to Protocol | 7 | 14
Not completed — Familial and Personal Reasons | 9 | 34
Not completed — Sponsor Decision | 4 | 10

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized patients who were exposed to at least 1 dose of study drug, regardless of the amount of treatment administered.The one patient in the placebo group who received Lixisenatide was described in the Lixisenatide group.
Groups:
- Placebo: 2-step initiation regimen of volume matching placebo: 10 mcg QD subcutaneously for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to the end of treatment.
- Total: Total of all reporting groups
Arm/Group | Placebo | Lixisenatide | Total
Number analyzed (Participants) | 285 | 574 | 859
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (10.1) | 57.0 (9.8) | 57.2 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 290 | 425
  Male | 150 | 284 | 434
Race/Ethnicity, Customized [Number; unit: participants]
  Race: Caucasian/White | 151 | 297 | 448
  Race: Black | 9 | 17 | 26
  Race: Asian/Oriental | 125 | 260 | 385
  Ethnicity: Hispanic | 5 | 18 | 23
  Ethnicity: Non Hispanic | 280 | 556 | 836
Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of hemoglobin] | 8.21 (0.84) | 8.28 (0.86) | 8.25 (0.85)
2-Hour Postprandial Plasma Glucose (PPG) [Mean (Standard Deviation); unit: millimole per liter (mmol/L)] — The 2-hour PPG test measured blood glucose 2 hours after eating a standardized meal. Number of patients analyzed = 154 and 309 for Placebo and Lixisenatide treatment arms, respectively.
  millimole per liter (mmol/L) | 16.44 (3.74) | 16.69 (4.02) | 16.60 (3.92)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 9.29 (2.37) | 9.67 (2.24) | 9.55 (2.29)
Body Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 84.42 (22.83) | 82.30 (21.76) | 83.00 (22.13)
Homeostasis Model Assessment for Beta-cell Function (HOMA-beta) [Mean (Standard Deviation); unit: percentage of normal beta cells function] — Beta cell function was assessed by HOMA-beta. HOMA-beta (percentage [%] of normal beta cells function) = (20 multiplied by fasting plasma insulin [micro unit per milliliter]) divided by (FPG [mmol/L] minus 3.5). Number of patients analyzed = 152 and 306 for Placebo and Lixisenatide treatment arms, respectively.
  percentage of normal beta cells function | 36.43 (39.43) | 34.28 (69.82) | 34.99 (61.39)
Fasting glucagon [Mean (Standard Deviation); unit: nanogram per liter (ng/L)] — Number of patients analyzed = 152 and 309 for Placebo and Lixisenatide treatment arm, respectively.
  nanogram per liter (ng/L) | 0.89 (0.55) | 0.83 (0.43) | 0.85 (0.47)
2-hour postprandial glucagon [Mean (Standard Deviation); unit: ng/L] — Number of patients analyzed = 149 and 300 for Placebo and Lixisenatide treatment arm, respectively.
  ng/L | 102.27 (39.37) | 97.83 (31.94) | 99.31 (34.60)
Fasting plasma insulin (FPI) [Mean (Standard Deviation); unit: picomole per liter (pmol/L)] — Number of patients analyzed = 152 and 306 for Placebo and Lixisenatide treatment arm, respectively.
  picomole per liter (pmol/L) | 66.89 (63.92) | 61.34 (52.63) | 63.18 (56.61)
2-hour postprandial plasma insulin [Mean (Standard Deviation); unit: pmol/L] — Number of patients analyzed = 154 and 305 for Placebo and Lixisenatide treatment arm, respectively.
  pmol/L | 281.26 (243.56) | 259.44 (182.64) | 266.76 (205.09)
Fasting proinsulin [Mean (Standard Deviation); unit: pmol/L] — Number of patients analyzed = 138 and 290 for Placebo and Lixisenatide treatment arm, respectively.
  pmol/L | 34.39 (32.61) | 33.35 (27.43) | 33.69 (29.17)
2-hour postprandial proinsulin [Mean (Standard Deviation); unit: pmol/L] — Number of patients analyzed = 130 and 257 for Placebo and Lixisenatide treatment arm, respectively.
  pmol/L | 61.73 (46.48) | 62.12 (44.80) | 61.99 (45.31)
Fasting C-peptide [Mean (Standard Deviation); unit: mmol/L] — Number of patients analyzed = 152 and 309 for Placebo and Lixisenatide treatment arm, respectively.
  mmol/L | 0.89 (0.55) | 0.83 (0.43) | 0.85 (0.47)
2-hour postprandial C-peptide [Mean (Standard Deviation); unit: mmol/L] — Number of patients analyzed = 152 and 308 for Placebo and Lixisenatide treatment arm, respectively.
  mmol/L | 2.12 (1.05) | 1.99 (0.90) | 2.03 (0.95)
Glucose Excursion [Mean (Standard Deviation); unit: mmol/L] — Glucose excursion = 2-hour PPG minus plasma glucose 30 minutes prior to the meal test, before study drug administration. Number of patients analyzed = 154 and 309 for Placebo and Lixisenatide treatment arms, respectively.
  mmol/L | 6.84 (3.78) | 6.99 (3.71) | 6.94 (3.73)
Fasting proinsulin-to-insulin ratio [Mean (Standard Deviation); unit: ratio] — Number of patients analyzed = 137 and 285 for Placebo and Lixisenatide treatment arm, respectively.
  ratio | 0.62 (0.36) | 0.70 (0.57) | 0.67 (0.51)
2-hour postprandial proinsulin-to-insulin ratio [Mean (Standard Deviation); unit: ratio] — Number of patients analyzed = 130 and 253 for Placebo and Lixisenatide treatment arm, respectively.
  ratio | 0.30 (0.22) | 0.32 (0.24) | 0.31 (0.23)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 24
Description: Absolute change = HbA1c value at Week 24 minus HbA1c value at baseline. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to 3 days after the last dose of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy. For a patient to be included in Modified Intent-to-Treat (mITT) population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population:all randomized patients who received at least 1 dose;had baseline,at least 1 post-baseline efficacy assessment, irrespective of compliance with study protocol/procedures. Last observation carried forward used. Number of patients analyzed=patients with baseline and at least 1 post-baseline HbA1c assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: percentage of hemoglobin
Groups:
- Placebo: 2-step initiation regimen of volume matching placebo.
- Lixisenatide: 2-step initiation regimen of lixisenatide.
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 274 | 544
percentage of hemoglobin | -0.10 (0.071) | -0.85 (0.061)
Statistical Analysis 1: Comparison: Placebo vs Lixisenatide; To detect a difference of 0.5% (or 0.4%) in change from baseline to Week 24 in HbA1c between lixisenatide and placebo, 570 patients in lixisenatide arm and 285 in placebo arm would provide a power of 99% (or 98%) assuming common standard deviation of 1.3% with a 2-sided test at 5% significance level; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing: 2-sided at significance level=0.05. Analysis of co-variance (ANCOVA) included treatment arms, randomization strata of screening HbA1c (<8.0, >=8.0%), metformin use (yes, no), country as fixed effects, baseline HbA1c as covariate; Least squares (LS) mean difference = -0.74, 95% CI 2-sided [-0.867 to -0.621], Standard Error of Mean 0.063

2. Secondary Outcome: Change From Baseline in 2-Hour Postprandial Plasma Glucose (PPG) at Week 24
Description: The 2-hour PPG blood sample was drawn 2 hours after start of a standardized meal (standardized meal challenge test performed in selected sites). Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to last dosing day of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: Subgroup for standardized meal test in mITT population. Missing data was imputed using last observation carried forward (LOCF). Here, number of patients analyzed = patients with baseline and at least 1 post-baseline 2-hour PPG assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 120 | 249
mmol/L | -0.21 (0.489) | -6.19 (0.408)

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to 1 day after the last dose of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline FPG assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 283 | 564
mmol/L | -0.36 (0.161) | -0.99 (0.139)

4. Secondary Outcome: Change From Baseline in Body Weight at Week 24
Description: Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to 3 days after the last dose of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline body weight assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: kilogram
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 278 | 554
kilogram | -0.93 (0.234) | -1.76 (0.202)

5. Secondary Outcome: Change From Baseline in Beta-cell Function Assessed by HOMA-beta at Week 24
Description: Beta cell function was assessed by HOMA-beta. HOMA-beta blood samples were drawn during a standardized meal challenge test (performed in selected sites). HOMA-beta (% of normal beta cells function) = (20 multiplied by fasting plasma insulin [micro unit per milliliter]) divided by (FPG [mmol/L] minus 3.5). Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to last dosing day of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: Subgroup for standardized meal test in mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline HOMA-beta assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: % of normal beta cells function
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 116 | 241
% of normal beta cells function | 6.63 (5.663) | 4.83 (4.686)

6. Other Pre Specified Outcome: Change From Baseline in Glucose Excursion at Week 24
Description: Glucose excursion = 2-hour PPG minus plasma glucose 30 minutes prior to the standardized meal test (performed in selected sites), before study drug administration. Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to last dosing day of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: Subgroup for standardized meal test in mITT population. Missing data was imputed using last observation carried forward (LOCF). Here, number of patients analyzed = patients with baseline and at least 1 post-baseline glucose excursion assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 120 | 249
mmol/L | 0.35 (0.432) | -5.22 (0.360)

7. Secondary Outcome: Change From Baseline in Fasting Glucagon and 2-hour Postprandial Glucagon at Week 24
Description: The fasting glucagon and the 2-hour postprandial glucagon blood samples were drawn during a standardized meal challenge test (performed in selected sites). Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to last dosing day of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: Subgroup for standardized meal test in mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline glucagon assessment during on-treatment period and 'n' = patients with baseline and at least 1 post-baseline assessment for the specified category.
Measure: Least Squares Mean (Standard Error); unit: ng/L
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 114 | 238
ng/L
  Fasting glucagon (n=111, 238) | 2.03 (2.566) | -2.10 (2.081)
  2-hour postprandial glucagon (n=114, 234) | -1.19 (2.999) | -23.33 (2.500)

8. Secondary Outcome: Change From Baseline in Fasting Plasma Insulin (FPI) and 2-hour Postprandial Plasma Insulin at Week 24
Description: The fasting plasma insulin and the 2-hour postprandial plasma insulin blood samples were drawn during a standardized meal challenge test (performed in selected sites). Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to last dosing day of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: Subgroup for standardized meal test in mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline plasma insulin assessment during on-treatment period and 'n' = patients with baseline and at least 1 post-baseline assessment for the specified category.
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 120 | 244
pmol/L
  FPI (n=117, 242) | 1.42 (6.587) | -4.03 (5.445)
  2-hour postprandial plasma insulin (n=120, 244) | -2.22 (18.754) | -67.67 (15.944)

9. Secondary Outcome: Change From Baseline in Fasting Proinsulin and 2-hour Postprandial Proinsulin at Week 24
Description: The fasting Proinsulin and the 2-hour postprandial Proinsulin blood samples were drawn during a standardized meal challenge test (performed in selected sites). Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to last dosing day of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: Subgroup for standardized meal test in mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline proinsulin assessment during on-treatment period and 'n' = patients with baseline and at least 1 post-baseline assessment for the specified category.
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 97 | 205
pmol/L
  Fasting proinsulin (n=97, 205) | -1.05 (1.983) | -6.33 (1.671)
  2-hour postprandial proinsulin (n=93, 193) | 3.55 (4.200) | -4.20 (3.550)

10. Other Pre Specified Outcome: Change From Baseline in Fasting Proinsulin-to-insulin Ratio and 2-hour Postprandial Proinsulin-to-insulin Ratio at Week 24
Description: The fasting proinsulin-to-insulin ratio and 2-hour postprandial proinsulin-to-insulin ratio were measured during a standardized meal challenge test (performed in selected sites). Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to last dosing day of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: Subgroup for standardized meal test in mITT population. Missing data imputed using LOCF. Number of patients analyzed=patients with baseline and at least 1 post-baseline proinsulin-to-insulin ratio assessment during on-treatment period and 'n'= patients with baseline and at least 1 post-baseline assessment for the specific category.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 95 | 199
ratio
  Fasting proinsulin-to-insulin ratio (n=95, 199) | -0.04 (0.049) | -0.13 (0.043)
  2-hour postprandial ratio (n=92, 190) | 0.01 (0.060) | 0.16 (0.053)

11. Secondary Outcome: Change From Baseline in Fasting C-peptide and 2-hour Postprandial C-peptide at Week 24
Description: The fasting C-peptide and the 2-hour postprandial C-peptide blood samples were drawn during a standardized meal challenge test (performed in selected sites). Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to last dosing day of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy.For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: Subgroup for standardized meal test in mITT population. Missing data was imputed using LOCF. here. number of patients analyzed = patients with baseline and at least 1 post-baseline C-peptide assessment during on-treatment period and 'n' = patients with baseline and at least 1 post-baseline assessment for the specified category.
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 119 | 248
nmol/L
  Fasting C-peptide (n=117, 244) | -0.06 (0.038) | -0.07 (0.031)
  2-hour postprandial C-peptide (n=119, 248) | -0.14 (0.087) | -0.37 (0.072)

12. Secondary Outcome: Percentage of Patients With Glycosylated Hemoglobin (HbA1c) Level Less Than 7% at Week 24
Description: The on-treatment period for this efficacy variable is time from the first dose of study drug and up to 3 days after the last dose of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Week 24
Population: mITT population. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline HbA1c assessment during on-treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 274 | 544
percentage of participants | 13.5 | 36.4

13. Secondary Outcome: Percentage of Patients With Glycosylated Hemoglobin (HbA1c) Level Less Than or Equal to 6.5% at Week 24
Description: as for outcome 12
Time Frame: Week 24
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 274 | 544
percentage of participants | 4.7 | 19.3

14. Other Pre Specified Outcome: Percentage of Patients With at Least 5% Weight Loss From Baseline at Week 24
Description: as for outcome 12
Time Frame: Baseline, Week 24
Population: mITT population. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline body weight assessment during on-treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 278 | 554
percentage of participants | 7.2 | 14.4

15. Secondary Outcome: Percentage of Patients Requiring Rescue Therapy During Main 24-Week Period
Description: Routine fasting self-monitored plasma glucose (SMPG) and central laboratory FPG (and HbA1c after week 12) values were used to determine the requirement of rescue medication. If fasting SMPG value exceeded the specified limit for 3 consecutive days, the central laboratory FPG (and HbA1c after week 12) were performed. Threshold values - from baseline to Week 8: fasting SMPG/FPG >270 milligram/deciliter (mg/dL) (15.0 mmol/L), from Week 8 to Week 12: fasting SMPG/FPG >240 mg/dL (13.3 mmol/L), and from Week 12 to Week 24: fasting SMPG/FPG >200 mg/dL (11.1 mmol/L) or HbA1c >8.5%. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline up to Week 24
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 286 | 570
percentage of participants | 12.6 | 4.0

16. Other Pre Specified Outcome: Number of Patients With Symptomatic Hypoglycemia and Severe Symptomatic Hypoglycemia
Description: Symptomatic hypoglycemia was an event with clinical symptoms that were considered to result from a hypoglycemic episode with an accompanying plasma glucose less than 60 mg/dL (3.3 mmol/L) or associated with prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration if no plasma glucose measurement was available. Severe symptomatic hypoglycemia was symptomatic hypoglycemia event in which the patient required the assistance of another person and was associated with either a plasma glucose level below 36 mg/dL (2.0 mmol/L) or prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration, if no plasma glucose measurement was available.
Time Frame: First dose of study drug up to 3 days after the last dose administration, for up to 120 weeks
Population: Safety population included all randomized patients who were exposed to at least 1 dose of study drug, regardless of the amount of treatment administered.The one patient in the placebo group who received Lixisenatide was analyzed in the Lixisenatide group
Measure: Number; unit: participants
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 285 | 574
participants
  Symptomatic hypoglycemia | 51 | 127
  Severe symptomatic hypoglycemia | 1 | 2

ADVERSE EVENTS:
Time Frame: First dose of study drug up to 3 days after the last dose administration, for up to 120 weeks
Description: Median exposure to study treatment was 617 and 610 days in placebo and lixisenatide treatment arms, respectively. The analysis was performed on safety population, defined as all randomized patients who were exposed to at least 1 dose of study drug, regardless of the amount of treatment administered. The one patient in the placebo group who received Lixisenatide was analyzed in the Lixisenatide group
Arm/Group | Placebo | Lixisenatide
Serious Adverse Events (participants affected / at risk) | 35/285 | 58/574
Other Adverse Events (participants affected / at risk) | 148/285 | 362/574
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=285) | Lixisenatide (N=574)
Arthritis bacterial (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0
Colitis herpes (Infections and infestations) | 1 | 0
Leptospirosis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 2
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glottis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Allergy to arthropod sting (Immune system disorders) | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Depression (Psychiatric disorders) | 0 | 1
Schizophrenia simple (Psychiatric disorders) | 0 | 1
Schizophrenia, paranoid type (Psychiatric disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 1 | 0
Essential tremor (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 1
Lacunar infarction (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 2
VIIth nerve paralysis (Nervous system disorders) | 1 | 1
Cataract (Eye disorders) | 0 | 1
Cataract nuclear (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 2
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 2
Angina pectoris (Cardiac disorders) | 2 | 1
Angina unstable (Cardiac disorders) | 1 | 2
Atrioventricular block complete (Cardiac disorders) | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 2
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 2
Aortic stenosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 1 | 0
Chest pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 0
Sudden cardiac death (General disorders) | 0 | 1
Blood calcitonin increased (Investigations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 3
Coronary angioplasty (Surgical and medical procedures) | 0 | 2
Coronary arterial stent insertion (Surgical and medical procedures) | 1 | 0
Percutaneous coronary intervention (Surgical and medical procedures) | 2 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=285) | Lixisenatide (N=574)
Influenza (Infections and infestations) | 11 | 30
Nasopharyngitis (Infections and infestations) | 58 | 91
Upper respiratory tract infection (Infections and infestations) | 21 | 43
Hypoglycaemia (Metabolism and nutrition disorders) | 55 | 140
Dizziness (Nervous system disorders) | 18 | 60
Headache (Nervous system disorders) | 20 | 44
Constipation (Gastrointestinal disorders) | 11 | 30
Diarrhoea (Gastrointestinal disorders) | 27 | 71
Dyspepsia (Gastrointestinal disorders) | 4 | 34
Nausea (Gastrointestinal disorders) | 25 | 161
Vomiting (Gastrointestinal disorders) | 15 | 61
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 36
Blood glucose decreased (Investigations) | 11 | 30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.